CLINICAL TRIAL: NCT00285337
Title: An Assessment of Surgical Techniques for Treating Cervical Spondylotic Myelopathy
Brief Title: Assessment of Surgical Techniques for Treating Cervical Spondylotic Myelopathy
Acronym: CSM
Status: Completed | Type: Observational
Sponsor: AOSpine North America Research Network (Network)
Collaborators: AOSpine North America (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-CSM-03
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Cervical Spondylotic Myelopathy
Keywords: Myelopathy; Laminectomy; Laminoplasty; Decompression of Spinal Cord; Cervical Spondylosis
MeSH Terms: conditions — Spinal Cord Diseases; Spondylosis | interventions — Laminectomy; Laminoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laminectomy and Laminoplasty — Posterior versus anterior approach to laminectomy and laminoplasty

SUMMARY:
The primary purpose of this study is to compare anterior and posterior surgical approach in treatment of CSM in terms of surgical complications and neurological, functional, disease-specific and quality of life outcomes measures.

Secondary aims are to quantify the amount of change pre and post-surgery concerning the same outcome measures; to determine if there are differences in outcomes between posterior surgical techniques (i.e. laminectomy with fusion or laminoplasty) and examine the relationship between baseline MRI and baseline and follow-up neurological and functional outcomes.

DETAILED DESCRIPTION:
Narrowing of the spinal canal by osteophytes, ossification of the posterior longitudinal ligament, or bulging of a large central disk can compress the cervical spinal cord and impinge the spinal nerve roots, resulting in neck pain and various degrees of neurological symptoms and impairment.2 In severe cases, this can lead to stenosis of the cervical spine, resulting in upper motor neuron symptoms in the lower extremity and lower motor neuron symptoms in the upper extremity. When conservative measures such as traction, cervical collar, and postural exercises fail to prevent neurologic progression, surgery may be indicated.

A variety of surgical approaches and procedures are available, and the optimal choice of treatment remains controversial. Surgical procedures designed to decompress the spinal cord and, in some cases, stabilize the spine have been shown to be successful, but there is a persistent percentage of patients who do not improve with surgical intervention.3 Additionally, the potential complications of surgery for CSM may depend on the various methods of surgical management. Historically, cervical laminectomy, a posterior approach, had been regarded as the standard surgical treatment of CSM. However, over the past 20 years, it has been increasingly recognized that laminectomy without fusion is not appropriate for all patients and may result in instability and deformity. Because of the instability caused by laminectomies, alternate surgical approaches such as anterior approaches to the spine and laminoplasty have been developed, and have gained increasing popularity over the years.3 A range of factors must be considered when deciding which surgical technique to use. Surgeons are often challenged with determining the most appropriate technique because there is limited information about whether there is a difference between surgical procedures in terms of clinical and radiographic outcomes, in postoperative complication rates and in functional and quality of life outcomes. Methods of treatment include conservative and surgical management. Among surgically managed patients, an anterior or posterior approach may be employed. Among those managed posteriorly, laminoplasty or laminectomy with fusion are common surgical techniques. With several standards of care available for this population, a better understanding of the corresponding positive and negative outcomes with respect to clinical and patient-centered outcomes is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo surgery for symptomatic cervical spondylotic myelopathy with one or or more of the following symptoms: Numb clumsy hands, impairment of gait, bilateral arm parasthesia, L'Hermitte's phenomena
* and one or more of the following signs: corticospinal distribution motor deficits, athropy of hand intrinsic muscles, hyperflexia, positive Hoffman sign, upgoing plantar responses, lower limb spasticity, broad based unstable gait

Exclusion Criteria:

* Asymptomatic cervical spondylotic myelopathy
* previous surgery for CSM
* Active infection
* Neoplastic disease
* Rheumatoid arthritis
* Ankylosing spondylitis
* Trauma
* Concomitant lumbar stenosis
* Not referred for surgical consultation
* Participating in other trials or unlikely to attend follow-ups

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2005-12; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Clinical and radiological outcomes, functional status and general health related quality of life between anterior vs. posterior approach | 12 months
Compare the rate of complications between operative patients managed with anterior vs. posterior approaches 6,12 and 24 months following surgery | 24 months

SECONDARY OUTCOMES:
Compare the outcome of operative treatment at baseline and 6, 12 and 24 months using Nurick score, 30m walk test, mJOA score, NDI and SF-36 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fehlings, MD, PhD, Principal Investigator — University of Toronto
Locations (13):
- United States (12):
  - Spine Education and Research Institute, Thornton, Colorado
  - Emory University, Atlanta, Georgia
  - Indianda Spine Group, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - New England Baptist Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Thomas Jefferson University and Rothman Institure Orthopaedics, Philadelphia, Pennsylvania
  - Universty of Utah, Salt Lake City, Utah
  - University Of Virginia, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Fehlings MG, Smith JS, Kopjar B, Arnold PM, Yoon ST, Vaccaro AR, Brodke DS, Janssen ME, Chapman JR, Sasso RC, Woodard EJ, Banco RJ, Massicotte EM, Dekutoski MB, Gokaslan ZL, Bono CM, Shaffrey CI. Perioperative and delayed complications associated with the surgical treatment of cervical spondylotic myelopathy based on 302 patients from the AOSpine North America Cervical Spondylotic Myelopathy Study. J Neurosurg Spine. 2012 May;16(5):425-32. doi: 10.3171/2012.1.SPINE11467. Epub 2012 Feb 10. PMID 22324802
- [Background] Fehlings MG, Jha NK, Hewson SM, Massicotte EM, Kopjar B, Kalsi-Ryan S. Is surgery for cervical spondylotic myelopathy cost-effective? A cost-utility analysis based on data from the AOSpine North America prospective CSM study. J Neurosurg Spine. 2012 Sep;17(1 Suppl):89-93. doi: 10.3171/2012.6.AOSPINE111069. PMID 22985375
- [Background] Karadimas SK, Gatzounis G, Fehlings MG. Pathobiology of cervical spondylotic myelopathy. Eur Spine J. 2015 Apr;24 Suppl 2:132-8. doi: 10.1007/s00586-014-3264-4. Epub 2014 Mar 14. PMID 24626958
- [Background] Wilson JR, Fehlings MG, Kalsi-Ryan S, Shamji MF, Tetreault LA, Rhee JM, Chapman JR. Diagnosis, heritability, and outcome assessment in cervical myelopathy: a consensus statement. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S76-7. doi: 10.1097/BRS.0b013e3182a7f4bf. PMID 23963010
- [Background] Fehlings MG, Wilson JR, Yoon ST, Rhee JM, Shamji MF, Lawrence BD. Symptomatic progression of cervical myelopathy and the role of nonsurgical management: a consensus statement. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S19-20. doi: 10.1097/BRS.0b013e3182a7f4de. PMID 23963011
- [Background] Kalsi-Ryan S, Karadimas SK, Fehlings MG. Cervical spondylotic myelopathy: the clinical phenomenon and the current pathobiology of an increasingly prevalent and devastating disorder. Neuroscientist. 2013 Aug;19(4):409-21. doi: 10.1177/1073858412467377. Epub 2012 Nov 30. PMID 23204243
- [Background] Shamji MF, Ames CP, Smith JS, Rhee JM, Chapman JR, Fehlings MG. Myelopathy and spinal deformity: relevance of spinal alignment in planning surgical intervention for degenerative cervical myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S147-8. doi: 10.1097/BRS.0b013e3182a7f521. PMID 23963013
- [Background] Lawrence BD, Shamji MF, Traynelis VC, Yoon ST, Rhee JM, Chapman JR, Brodke DS, Fehlings MG. Surgical management of degenerative cervical myelopathy: a consensus statement. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S171-2. doi: 10.1097/BRS.0b013e3182a7f4ff. PMID 23963012
- [Background] Liu S, Lafage R, Smith JS, Protopsaltis TS, Lafage VC, Challier V, Shaffrey CI, Radcliff K, Arnold PM, Chapman JR, Schwab FJ, Massicotte EM, Yoon ST, Fehlings MG, Ames CP. Impact of dynamic alignment, motion, and center of rotation on myelopathy grade and regional disability in cervical spondylotic myelopathy. J Neurosurg Spine. 2015 Dec;23(6):690-700. doi: 10.3171/2015.2.SPINE14414. Epub 2015 Aug 28. PMID 26315953
- [Result] Arnold PM, Fehlings MG, Kopjar B, Yoon ST, Massicotte EM, Vaccaro AR, Brodke DS, Shaffrey CI, Smith JS, Woodard EJ, Banco RJ, Chapman JR, Janssen ME, Bono CM, Sasso RC, Dekutoski MB, Gokaslan ZL. Mild diabetes is not a contraindication for surgical decompression in cervical spondylotic myelopathy: results of the AOSpine North America multicenter prospective study (CSM). Spine J. 2014 Jan;14(1):65-72. doi: 10.1016/j.spinee.2013.06.016. Epub 2013 Aug 24. PMID 23981820
- [Result] Fehlings MG, Wilson JR, Kopjar B, Yoon ST, Arnold PM, Massicotte EM, Vaccaro AR, Brodke DS, Shaffrey CI, Smith JS, Woodard EJ, Banco RJ, Chapman JR, Janssen ME, Bono CM, Sasso RC, Dekutoski MB, Gokaslan ZL. Efficacy and safety of surgical decompression in patients with cervical spondylotic myelopathy: results of the AOSpine North America prospective multi-center study. J Bone Joint Surg Am. 2013 Sep 18;95(18):1651-8. doi: 10.2106/JBJS.L.00589. PMID 24048552
- [Result] Tetreault LA, Kopjar B, Vaccaro A, Yoon ST, Arnold PM, Massicotte EM, Fehlings MG. A clinical prediction model to determine outcomes in patients with cervical spondylotic myelopathy undergoing surgical treatment: data from the prospective, multi-center AOSpine North America study. J Bone Joint Surg Am. 2013 Sep 18;95(18):1659-66. doi: 10.2106/JBJS.L.01323. PMID 24048553
- [Result] Karpova A, Arun R, Kalsi-Ryan S, Massicotte EM, Kopjar B, Fehlings MG. Do quantitative magnetic resonance imaging parameters correlate with the clinical presentation and functional outcomes after surgery in cervical spondylotic myelopathy? A prospective multicenter study. Spine (Phila Pa 1976). 2014 Aug 15;39(18):1488-97. doi: 10.1097/BRS.0000000000000436. PMID 24859570
- [Result] Fehlings MG, Barry S, Kopjar B, Yoon ST, Arnold P, Massicotte EM, Vaccaro A, Brodke DS, Shaffrey C, Smith JS, Woodard E, Banco RJ, Chapman J, Janssen M, Bono C, Sasso R, Dekutoski M, Gokaslan ZL. Anterior versus posterior surgical approaches to treat cervical spondylotic myelopathy: outcomes of the prospective multicenter AOSpine North America CSM study in 264 patients. Spine (Phila Pa 1976). 2013 Dec 15;38(26):2247-52. doi: 10.1097/BRS.0000000000000047. PMID 24108289
- [Result] Kopjar B, Tetreault L, Kalsi-Ryan S, Fehlings M. Psychometric properties of the modified Japanese Orthopaedic Association scale in patients with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2015 Jan 1;40(1):E23-8. doi: 10.1097/BRS.0000000000000648. PMID 25341993
- [Result] Arvin B, Kalsi-Ryan S, Karpova A, Mercier D, Furlan JC, Massicotte EM, Fehlings MG. Postoperative magnetic resonance imaging can predict neurological recovery after surgery for cervical spondylotic myelopathy: a prospective study with blinded assessments. Neurosurgery. 2011 Aug;69(2):362-8. doi: 10.1227/NEU.0b013e31821a418c. PMID 21471834
- [Result] Furlan JC, Kalsi-Ryan S, Kailaya-Vasan A, Massicotte EM, Fehlings MG. Functional and clinical outcomes following surgical treatment in patients with cervical spondylotic myelopathy: a prospective study of 81 cases. J Neurosurg Spine. 2011 Mar;14(3):348-55. doi: 10.3171/2010.10.SPINE091029. Epub 2011 Jan 14. PMID 21235299
- [Result] Singh A, Tetreault L, Fehlings MG, Fischer DJ, Skelly AC. Risk factors for development of cervical spondylotic myelopathy: results of a systematic review. Evid Based Spine Care J. 2012 Aug;3(3):35-42. doi: 10.1055/s-0032-1327808. PMID 23526904
- [Result] Skelly AC, Hashimoto RE, Norvell DC, Dettori JR, Fischer DJ, Wilson JR, Tetreault LA, Fehlings MG. Cervical spondylotic myelopathy: methodological approaches to evaluate the literature and establish best evidence. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S9-18. doi: 10.1097/BRS.0b013e3182a7ebbf. PMID 24026148
- [Result] Yoon ST, Raich A, Hashimoto RE, Riew KD, Shaffrey CI, Rhee JM, Tetreault LA, Skelly AC, Fehlings MG. Predictive factors affecting outcome after cervical laminoplasty. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S232-52. doi: 10.1097/BRS.0b013e3182a7eb55. PMID 23962999
- [Result] Fehlings MG, Tetreault LA, Wilson JR, Skelly AC. Cervical spondylotic myelopathy: current state of the art and future directions. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S1-8. doi: 10.1097/BRS.0b013e3182a7e9e0. PMID 23962994
- [Result] Kalsi-Ryan S, Singh A, Massicotte EM, Arnold PM, Brodke DS, Norvell DC, Hermsmeyer JT, Fehlings MG. Ancillary outcome measures for assessment of individuals with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S111-22. doi: 10.1097/BRS.0b013e3182a7f499. PMID 23963009
- [Result] Shamji MF, Massicotte EM, Traynelis VC, Norvell DC, Hermsmeyer JT, Fehlings MG. Comparison of anterior surgical options for the treatment of multilevel cervical spondylotic myelopathy: a systematic review. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S195-209. doi: 10.1097/BRS.0b013e3182a7eb27. PMID 23962998
- [Result] Smith JS, Lafage V, Ryan DJ, Shaffrey CI, Schwab FJ, Patel AA, Brodke DS, Arnold PM, Riew KD, Traynelis VC, Radcliff K, Vaccaro AR, Fehlings MG, Ames CP. Association of myelopathy scores with cervical sagittal balance and normalized spinal cord volume: analysis of 56 preoperative cases from the AOSpine North America Myelopathy study. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S161-70. doi: 10.1097/BRS.0b013e3182a7eb9e. PMID 23963001
- [Result] Karadimas SK, Erwin WM, Ely CG, Dettori JR, Fehlings MG. Pathophysiology and natural history of cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S21-36. doi: 10.1097/BRS.0b013e3182a7f2c3. PMID 23963004
- [Result] Karpova A, Arun R, Davis AM, Kulkarni AV, Massicotte EM, Mikulis DJ, Lubina ZI, Fehlings MG. Predictors of surgical outcome in cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Mar 1;38(5):392-400. doi: 10.1097/BRS.0b013e3182715bc3. PMID 23448898
- [Result] Karpova A, Arun R, Davis AM, Kulkarni AV, Mikulis DJ, Sooyong C, Rabin D, Craciunas S, Smith SR, Hansen MA, George J, Fehlings MG. Reliability of quantitative magnetic resonance imaging methods in the assessment of spinal canal stenosis and cord compression in cervical myelopathy. Spine (Phila Pa 1976). 2013 Feb 1;38(3):245-52. doi: 10.1097/BRS.0b013e3182672307. PMID 22772577
- [Result] Karpova A, Arun R, Cadotte DW, Davis AM, Kulkarni AV, O'Higgins M, Fehlings MG. Assessment of spinal cord compression by magnetic resonance imaging--can it predict surgical outcomes in degenerative compressive myelopathy? A systematic review. Spine (Phila Pa 1976). 2013 Jul 15;38(16):1409-21. doi: 10.1097/BRS.0b013e31829609a0. PMID 23591658
- [Result] Tetreault LA, Dettori JR, Wilson JR, Singh A, Nouri A, Fehlings MG, Brodt ED, Jacobs WB. Systematic review of magnetic resonance imaging characteristics that affect treatment decision making and predict clinical outcome in patients with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S89-110. doi: 10.1097/BRS.0b013e3182a7eae0. PMID 23962996
- [Result] Tetreault L, Nouri A, Singh A, Fawcett M, Nater A, Fehlings MG. An Assessment of the Key Predictors of Perioperative Complications in Patients with Cervical Spondylotic Myelopathy Undergoing Surgical Treatment: Results from a Survey of 916 AOSpine International Members. World Neurosurg. 2015 May;83(5):679-90. doi: 10.1016/j.wneu.2015.01.021. Epub 2015 Feb 12. PMID 25681596
- [Result] Tetreault LA, Cote P, Kopjar B, Arnold P, Fehlings MG; AOSpine North America and International Clinical Trial Research Network. A clinical prediction model to assess surgical outcome in patients with cervical spondylotic myelopathy: internal and external validations using the prospective multicenter AOSpine North American and international datasets of 743 patients. Spine J. 2015 Mar 1;15(3):388-97. doi: 10.1016/j.spinee.2014.12.145. Epub 2014 Dec 27. PMID 25549860
- [Result] Tetreault LA, Karpova A, Fehlings MG. Predictors of outcome in patients with degenerative cervical spondylotic myelopathy undergoing surgical treatment: results of a systematic review. Eur Spine J. 2015 Apr;24 Suppl 2:236-51. doi: 10.1007/s00586-013-2658-z. Epub 2013 Feb 6. PMID 23386279
- [Result] Mohanty C, Massicotte EM, Fehlings MG, Shamji MF. Association of preoperative cervical spine alignment with spinal cord magnetic resonance imaging hyperintensity and myelopathy severity: analysis of a series of 124 cases. Spine (Phila Pa 1976). 2015 Jan 1;40(1):11-6. doi: 10.1097/BRS.0000000000000670. PMID 25341991
- [Result] Nouri A, Tetreault L, Cote P, Zamorano JJ, Dalzell K, Fehlings MG. Does Magnetic Resonance Imaging Improve the Predictive Performance of a Validated Clinical Prediction Rule Developed to Evaluate Surgical Outcome in Patients With Degenerative Cervical Myelopathy? Spine (Phila Pa 1976). 2015 Jul 15;40(14):1092-100. doi: 10.1097/BRS.0000000000000919. PMID 25893357
- [Result] Nouri A, Tetreault L, Singh A, Karadimas SK, Fehlings MG. Degenerative Cervical Myelopathy: Epidemiology, Genetics, and Pathogenesis. Spine (Phila Pa 1976). 2015 Jun 15;40(12):E675-93. doi: 10.1097/BRS.0000000000000913. PMID 25839387
- [Result] Nouri A, Tetreault L, Zamorano JJ, Dalzell K, Davis AM, Mikulis D, Yee A, Fehlings MG. Role of magnetic resonance imaging in predicting surgical outcome in patients with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2015 Feb 1;40(3):171-8. doi: 10.1097/BRS.0000000000000678. PMID 25668335
- [Result] Singh A, Tetreault L, Casey A, Laing R, Statham P, Fehlings MG. A summary of assessment tools for patients suffering from cervical spondylotic myelopathy: a systematic review on validity, reliability and responsiveness. Eur Spine J. 2015 Apr;24 Suppl 2:209-28. doi: 10.1007/s00586-013-2935-x. Epub 2013 Sep 5. PMID 24005994
- [Result] Liu S, Tetreault L, Fehlings MG, Challier V, Smith JS, Shaffrey CI, Arnold PM, Scheer JK, Chapman JR, Kopjar B, Protopsaltis TS, Lafage V, Schwab F, Massicotte EM, Yoon ST, Ames CP. Novel Method Using Baseline Normalization and Area Under the Curve to Evaluate Differences in Outcome Between Treatment Groups and Application to Patients With Cervical Spondylotic Myelopathy Undergoing Anterior Versus Posterior Surgery. Spine (Phila Pa 1976). 2015 Dec;40(24):E1299-304. doi: 10.1097/BRS.0000000000001152. PMID 26335673
- [Derived] Bak AB, Moghaddamjou A, Arnold PM, Harrop JS, Fehlings MG. Chronic pain after decompression for degenerative cervical myelopathy: a pooled trajectory analysis of individual participant data. Pain. 2025 Oct 15. doi: 10.1097/j.pain.0000000000003828. Online ahead of print. PMID 41086299
- [Derived] Wong R, Alvi MA, Quddusi AI, Fehlings MG. Role of Neck Pain in Defining Clinical Trajectories of Outcomes in Patients With Degenerative Cervical Myelopathy: Results of a Novel Machine Learning Algorithm. Global Spine J. 2025 May 10;16(1):21925682251341263. doi: 10.1177/21925682251341263. Online ahead of print. PMID 40347099
- [Derived] Pedro KM, Alvi MA, Hejrati N, Moghaddamjou A, Fehlings MG. Elderly Patients Show Substantial Improvement in Health-Related Quality of Life After Surgery for Degenerative Cervical Myelopathy Despite Medical Frailty: An Ambispective Analysis of a Multicenter, International Data Set. Neurosurgery. 2024 Jan 10. doi: 10.1227/neu.0000000000002818. Online ahead of print. PMID 38197642
- [Derived] Merali ZG, Witiw CD, Badhiwala JH, Wilson JR, Fehlings MG. Using a machine learning approach to predict outcome after surgery for degenerative cervical myelopathy. PLoS One. 2019 Apr 4;14(4):e0215133. doi: 10.1371/journal.pone.0215133. eCollection 2019. PMID 30947300